CLINICAL TRIAL: NCT05451927
Title: A Randomized Double Blind Study to Examine the Effect of Natural Anti-obesity Agent Among Women of Lahore
Brief Title: Trial to Examine the Effect of Natural Anti- Obesity Agent (Phaseolus Vulgaris) Among Women of Lahore
Acronym: PVE-AO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hafiza Aisha Sadiqa (Other)
Collaborators: University of the Punjab (Other)
Responsible Party: Sponsor-Investigator, Hafiza Aisha Sadiqa, Student, University of the Punjab
Organization: University of the Punjab (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RCT012022
Record Dates: First submitted 2022-07-01; First posted 2022-07-11 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Overweight and Obesity
Keywords: Weight loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phaseolus Vulgaris (Experimental): Three oral doses of 1000 mg Phaseolus Vulgaris daily for 3 months
  Interventions: Dietary Supplement: Phaseolus Vulgaris
- Placebo (Placebo Comparator): Three oral doses of Placebo daily for 3 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Phaseolus Vulgaris — Weight loss
  Arms: Phaseolus Vulgaris
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This double-blind randomized placebo-controlled trial will test the hypothesis that administration of Phaseolus Vulgaris supplementation to women in Lahore, Pakistan, who are overweight will induce the weight loss (Primary outcome) and changes in body composition (Waist circumference) secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* BMI ranges from 25-40
* Consistently stable body weight for at least 6 months
* Good general health
* No ongoing drug treatment for weight reduction
* Commitment to avoid any changes in lifestyle throughout the test period
* Age between 18-45 years
* Women resident of Lahore

Exclusion Criteria:

* Pregnant or breast-feeding females
* People with Type 2 diabetes
* People with any other chronic diseases
* Weight reduction treatment during the 6 months prior to the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women, resident of Lahore, Pakistan
Enrollment: 72 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Body weight | 3 months
  change in body weight

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Sadiqa, M.Phil, Principal Investigator — University of the Punjab
Locations (2):
- Pakistan (2):
  - Akhuwat Medical Centre, Lahore, Punjab Province
  - Niazi Medical Centre, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared with other researchers subject to terms of Data Transfer Agreement and IRB approval
Supporting Information: CSR
Time Frame: Till 10 years after completion of trial
Access Criteria: on request through email and after Data Transfer Agreement and IRB approval